CLINICAL TRIAL: NCT03914521
Title: Pre-surgical CT Scan Assessment of Femoral Head Bone Mineral Density Before Resection of Neurogenic Heterotopic Ossification (NHO) of the Hip
Brief Title: Pre-surgical CT Scan Assessment of Bone Mineral Density Before Resection of NHO of the Hip
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0095
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Paraosteoarthropathies
Keywords: hip surgery; bone mineral density; femoral head; Pre-surgical prognostic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurogenic heterotopic ossification (NHO) is defined as an ectopic ossification around proximal joints usually seen after traumatic brain injury, spinal cord injury or polytrauma.

NHO causes pain, partial or total joint ankylosis and vascular or nerve complications.

The osteopenia (low bone density) induced by ankylose increases the fracture risk of femoral neck during the hip surgery performed to remove the NHO.

The analyse of femoral head bone mineral density from hip pre-surgical CT scan could anticipate this kind of complication establishing a presurgical prognostic.

If as it turns out the bone density measured from hip pre-surgical CT scan is relevant fracture risk marker, a preventive osteosynthesis or femoral head and neck resection could be performed in the same time of NHO resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients having surgery resection of surgery resection of Neurogenic heterotopic ossification of hip.
* Patients with pre-surgery CT-scan and surgery report available

Exclusion criteria:

* Minor patients
* Patients didn't have surgery surgery resection of Neurogenic heterotopic ossification of hip.
* Pre-surgery CT-scan and surgery report not available

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having surgery resection of surgery resection of Neurogenic heterotopic ossification of hip.
  Their per-operative CT-scan and surgery report will be collected from the records of Nîmes and Montpellier University Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
femoral head bone mineral density | 1 year
  femoral head bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Florence BAUMANN, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC